CLINICAL TRIAL: NCT03239743
Title: A Pilot Study to Evaluate the Efficacy of Virtual Reality on Pre-Operative Anxiety and Induction of Anesthesia in a Children's Hospital
Brief Title: Effects of Virtual Reality on Pre-Operative Anxiety and Induction of Anesthesia in Children and Adolescents
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Valley Anesthesiology Consultants (Other)
Collaborators: KindVR (Unknown); Phoenix Children's Hospital (Other)
Responsible Party: Principal Investigator, Neil Raj Singhal, Pain Management Research Director, Valley Anesthesiology Consultants
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17-025
Record Dates: First submitted 2017-04-21; First posted 2017-08-04 (Actual); Last update posted 2018-10-19 (Actual); Status verified 2018-10

CONDITIONS: Tonsillectomy
Keywords: virtual reality; adenoidectomy; induction of anesthesia; pre-operative anxiety
MeSH Terms: interventions — Midazolam

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Reality Group (Experimental): Subjects will be given the virtual reality device to interact with prior to surgery without the use of a pre-medication.
  Interventions: Device: Virtual Reality
- Midazolam Group (Active Comparator): Subjects will be given the drug Midazolam to help alleviate the pre-operative anxiety.
  Interventions: Drug: Midazolam

INTERVENTIONS:
Device: Virtual Reality — Child will wear and interact with virtual reality headset while waiting for surgery.
  Other Names: KindVR
  Arms: Virtual Reality Group
Drug: Midazolam — Child will receive Midazolam to help with pre-operative anxiety prior to surgery
  Other Names: Versed
  Arms: Midazolam Group

SUMMARY:
Pain and anxiety have a direct correlation. Patients who experience anxiety are more susceptible to feeling pain, and patients who experience pain are more likely to have a component of anxiety associated with their pain. A common technique used by pain psychologists to help minimize pain is distraction. Different forms of distraction include video games, movies, music, etc. Recently, doctors and researchers around the world have begun experimenting with Virtual Reality as a distraction technique.

A review of the use of virtual reality compared to the current standard of care may help uncover important trends regarding anxiety, postoperative pain and analgesic use in patients who undergo a tonsillectomy or a tonsillectomy and adenoidectomy.

DETAILED DESCRIPTION:
There are approximately five million pediatric surgeries performed in the United States every year, and approximately 50% of pediatric patients experience significant stress and anxiety before their surgery. High anxiety can result in increased postoperative pain, increased analgesic consumption, and delayed recovery. The perception of pain can have a strong psychological component and can increase if the patient gives the area of injury constant attention. Thus, different distraction techniques have been utilized by pain psychologists to take the patient's attention away from the area of injury.

Pharmacological intervention to treat preoperative anxiety in children has its own side-effect profile. Midazolam is a common medication used parentally, nasally, or orally to alleviate preoperative anxiety. However, there are many side-effects that are not always preventable. Reports of 3.8% of patients having paradoxical effects from midazolam have been documented, and delayed emergence is possible in surgeries of short duration. In addition, midazolam can also result in critical events perioperatively, such as airway obstruction and worsened nausea and vomiting. Non-pharmacological interventions could help avoid these complications, however, current studies do not show a viable alternative to a pharmacological interventions.

Virtual Reality (VR) is a technology that allows individuals to experience a virtual world. VR initially began as a form of entertainment, but it has expanded its application into several other areas. Within the past 10 years, this type of technology has been applied clinically as a method of distraction for medical procedures such as chemotherapy, physical therapy, burn wound changes, and surgery. VR allows the patients to be immersed in an interactive world stimulating sights, sounds, and motion to help enhance the distraction from pain, ultimately reducing anxiety. A small validation study was conducted at the Virtual Reality Medical Center to test the usability and safety in patients with chronic pain. Patients were presented with pleasant relaxing scenes including natural areas like forests, beaches, and mountains, with relaxing and soothing effects to help mimic slowed breathing. Researchers in this study found that the pain distraction virtual environment (VE) was easy to use, had good stereo sound effects, and was immersive and interactive. They also found that patients experienced low levels of fatigue, headache, eyestrain, and nausea when using the VR device. No studies have involved VR in setting of anesthesia induction period and a non-pharmacological intervention for preoperative anxiety.

A pilot study conducted by Wiederhold et al, tested 6 chronic pain patients using a head-mounted VR device. All six study participants reported a significant drop in pain while using the natural VE. Similarly, a study from the University of Washington found that children playing VR video games or navigating through a virtual environment while receiving wound care for their burns had lower pain scores than patients who just played video games. Another study conducted by Wiederhold et al., looked at fear and pain before and after dental treatment and found a significant decrease in pain perception and stated anxiety scores in patients using the VR eyeglasses compared to the nonuse group.

Based on success in other medical procedures, we propose a study to examine the efficacy and feasibility of using VR during induction of anesthesia to help minimize anxiety, postoperative pain and analgesic use in patients undergoing a tonsillectomy or a tonsillectomy and adenoidectomy procedure.

ELIGIBILITY:
Inclusion Criteria:

* Any patient undergoing tonsillectomy or tonsillectomy and adenoidectomy procedure
* Must be between the ages of 5 and 11 years
* Anxious/moderate anxiety patients (mYPAS greater than or equal to 30)

Exclusion Criteria:

* Any patient with preoperative peripherally placed IV
* Any patient who is cognitively impaired
* Any patient with a previous surgery
* ASA Physical Status higher than II
* Body Mass Index >30
* A history of affective disorder, attention disorder, or psychotropic medication use
* Calm/low anxiety patients (mYPAS less than 30)
* Deaf or blind

Ages: 5 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2017-07-20 (Actual); Primary Completion 2019-05 (Estimated); Study Completion 2019-05 (Estimated)

PRIMARY OUTCOMES:
Pre-Operative Anxiety measured by mYPAS anxiety scores | Baseline
  Determine if the use of a VR device will result in lower mYPAS anxiety scores during the preoperative period

SECONDARY OUTCOMES:
Induction Compliance of Anesthesia measured by the induction compliance checklist | Baseline
  Determine if the use of a VR device will result in greater induction of anesthesia measured by the induction compliance checklist.
Post-Operative Emergence Delirium measured by the PAED scale | up to 3 hours post operative
  Determine if VR use will reduce incidence of post-operative emergence delirium measured by the PAED scale.
Post-Operative Pain | up to 3 hours post operative
  Measure if VR use will reduce post-operative pain scores compared to patients receiving standard of care.
Post-Operative Opioid Use | up to 3 hours post operative
  Measure VR use will reduce opioid use compared to patients receiving standard of care

CONTACTS AND LOCATIONS:
Locations (1):
- Phoenix Children's Hospital, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mahrer NE, Gold JI. The use of virtual reality for pain control: a review. Curr Pain Headache Rep. 2009 Apr;13(2):100-9. doi: 10.1007/s11916-009-0019-8. PMID 19272275
- [Background] Wiederhold BK, Gao K, Sulea C, Wiederhold MD. Virtual reality as a distraction technique in chronic pain patients. Cyberpsychol Behav Soc Netw. 2014 Jun;17(6):346-52. doi: 10.1089/cyber.2014.0207. PMID 24892196
- [Background] Kain ZN, Mayes LC, Caldwell-Andrews AA, Karas DE, McClain BC. Preoperative anxiety, postoperative pain, and behavioral recovery in young children undergoing surgery. Pediatrics. 2006 Aug;118(2):651-8. doi: 10.1542/peds.2005-2920. PMID 16882820
- [Background] Kain ZN, Mayes LC, O'Connor TZ, Cicchetti DV. Preoperative anxiety in children. Predictors and outcomes. Arch Pediatr Adolesc Med. 1996 Dec;150(12):1238-45. doi: 10.1001/archpedi.1996.02170370016002. PMID 8953995
- [Background] Wiederhold MD, Gao K, Wiederhold BK. Clinical use of virtual reality distraction system to reduce anxiety and pain in dental procedures. Cyberpsychol Behav Soc Netw. 2014 Jun;17(6):359-65. doi: 10.1089/cyber.2014.0203. PMID 24892198
- [Background] Mosso-Vazquez JL, Gao K, Wiederhold BK, Wiederhold MD. Virtual reality for pain management in cardiac surgery. Cyberpsychol Behav Soc Netw. 2014 Jun;17(6):371-8. doi: 10.1089/cyber.2014.0198. PMID 24892200
- [Background] Wiederhold BK, Soomro A, Riva G, Wiederhold MD. Future directions: advances and implications of virtual environments designed for pain management. Cyberpsychol Behav Soc Netw. 2014 Jun;17(6):414-22. doi: 10.1089/cyber.2014.0197. PMID 24892206
- [Background] Hoffman HG, Chambers GT, Meyer WJ 3rd, Arceneaux LL, Russell WJ, Seibel EJ, Richards TL, Sharar SR, Patterson DR. Virtual reality as an adjunctive non-pharmacologic analgesic for acute burn pain during medical procedures. Ann Behav Med. 2011 Apr;41(2):183-91. doi: 10.1007/s12160-010-9248-7. PMID 21264690